CLINICAL TRIAL: NCT02358343
Title: ASCEND: A Trial of Sertraline vs. CBT for End-stage Renal Disease Patients With Depression
Brief Title: A Trial of Sertraline vs. CBT for End-stage Renal Disease Patients With Depression {ASCEND}
Acronym: ASCEND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: University of Texas (Other); University of New Mexico (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Rajnish Mehrotra, Professor of Medicine, Division of Nephrology, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 48647
Record Dates: First submitted 2015-01-13; First posted 2015-02-06 (Estimated); Results first posted 2019-07-23 (Actual); Last update posted 2019-07-23 (Actual); Status verified 2019-07

CONDITIONS: Depression; End Stage Renal Disease
Keywords: Comorbid Depression; Major Depressive Disorder; Dysthymia; Cognitive Behavioral therapy (CBT); Sertraline; Engagement Interview; End Stage Renal Disease (ESRD); Hemodialysis
MeSH Terms: conditions — Depression; Kidney Failure, Chronic; Depressive Disorder, Major; Dysthymic Disorder | interventions — Cognitive Behavioral Therapy; Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Engagement Interview (Active Comparator): Subjects will be randomly assigned to engagement interview or a control visit.Trained CBT therapists at each of the three sites will conduct the engagement interview. The session will be aimed at improving the acceptance of the diagnosis of depression by patients and treatment for the same.
  Interventions: Behavioral: Engagement Interview
- Control Visit (No Intervention): Subjects will be randomly assigned to engagement interview or a control visit. Individuals assigned to control visit will be scheduled for a follow-up discussion with a member of the research team. During this session, they will be informed of the diagnosis of major depression or dysthymia, the options for treatment available through the clinical trial, and alternatives should they decline participation in the clinical trial.
- Cognitive Behavioral Therapy (Active Comparator): The subjects will be randomly assigned to individual CBT or sertraline drug therapy using block randomization.
  Individuals will undergo 10 CBT sessions of 60 minutes each, by a trained therapist in the dialysis facility (8 weekly sessions; then every other week x 2). The CBT will be administered while the patient is undergoing HD; however, alternative arrangements will be made upon individual patient's preferences.
  Interventions: Behavioral: Cognitive Behavioral Therapy
- Antidepressant Drug Therapy (Active Comparator): The subjects will be randomly assigned to individual CBT or sertraline drug therapy using block randomization. Anti-Depressant Drug Therapy will be delivered with sertraline, a selective serotonin reuptake inhibitor, and the dose will be titrated using the Measurement Based Care Protocol.
  Interventions: Drug: Antidepressant Drug Therapy
- Observational Cohort (No Intervention): Subjects who (1) are not willing to participate in the clinical trial and (2) do not find any treatment acceptable outside the clinical trial will be invited to participate in the prospective observational cohort for serial assessment of depressive symptoms.These subjects will only undergo assessment of severity of depressive symptoms at weeks 0, 6, and 12 using QIDS-C.

INTERVENTIONS:
Behavioral: Engagement Interview — An Engagement Interview will comprise a one-on-one session with the patient, during which the health-care provider will use reflective statements and non-judgmental listening techniques, will explore barriers to treatment, and will help patient articulate ambivalence about engaging in treatment. This session will be enhanced with a 40-minute DVD that the subject will watch with the therapist in the dialysis facility. The subject will be encouraged to take the DVD home with them and watch it with their family members as well.
  Arms: Engagement Interview
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy (CBT) is a short-term psychotherapy that will focus on how the individual is thinking, behaving, and communicating today rather than on their childhood experience. The therapist will assist the patient in identifying specific distortions (cognitive assessment) and biases in thinking and will provide guidance on how to change this thinking. During the course of intervention, study subjects will undergo assessment of severity of depressive symptoms using Quick Inventory of Depressive Symptoms - Self-Report (QIDS-SR) every two weeks for the first six weeks (weeks 0, 2, 4, and 6) and every three weeks for the next six weeks (weeks 9 and 12).
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy
Drug: Antidepressant Drug Therapy — The site investigators will prescribe sertraline drug at a starting dose of 25 mg oral tablets. Dose titration will be implemented using standardized assessments of depressive symptoms and drug side effects; and the research team and the patient make joint decisions to maintain, increase, or decrease the dose. This will help establish the highest effective but tolerable dose tailored for each patient. The QIDS-SR scale will be used to assess the clinical response for dose titration. The FIBSER scale will be used to assess side effects and the degree to which they interfere with day-to-day functions. The participant-specific dose at week 6, up to a maximum of 200 mg/d, will be continued for the remaining 6 weeks.
  Other Names: Sertraline, "Zoloft"
  Arms: Antidepressant Drug Therapy

SUMMARY:
Patients whose kidneys fail generally require dialysis treatments to sustain life. The ability of patients to make major adjustments in their lives for dialysis is hampered by depression that affects almost one-quarter of such individuals. There are no studies that have adequately tested whether treatment of depression is effective in dialysis patients and if there is any difference between the response to the two most commonly available forms of treatment, psychotherapy and anti-depressant drug therapy.

To fill this important gap in the investigators knowledge, the investigators propose to undertake (1) a randomized controlled clinical trial of 200 patients to test whether an engagement interview will result in a higher proportion of dialysis patients accepting treatment for depression; and (2) a randomized controlled clinical trial of 120 patients to determine whether there is any difference in the likelihood of improvement of depressive symptoms with psychotherapy or drug therapy among dialysis patients with depression. Patients in these studies will be enrolled from among individuals receiving care in 50 dialysis facilities in three metropolitan areas - Seattle, Dallas, and Albuquerque. The research proposal has been developed with the support of patients, caregivers, and stakeholders to ensure that the findings from the study are relevant to them and can be readily implemented in day-to-day clinical practice. Hence, the engagement interview and psychotherapy will be delivered in a dialysis facility to ease the burden on patients, and the dose of the study drug will be changed in partnership with the study participants. In addition to depressive symptoms, the effect of treatment on other meaningful outcomes such as fatigue and sleep will be determined.

The two forms of treatment for depression being tested in this clinical trial are very different from each other and patients differ with regards to the treatment option preferable and/or available to them. Successful completion of the clinical trial will provide patients, caregivers, and other stakeholders with the information that they would need when faced with a diagnosis of depression in patients undergoing hemodialysis. This will allow patients to select evidence-based treatments to improve outcomes that are relevant to them.

DETAILED DESCRIPTION:
BACKGROUND Patients with end-stage renal disease undergoing maintenance hemodialysis (HD) have to adjust to complex treatment regimens, and experience frequent care transitions. This is compounded by a four-fold higher prevalence of comorbid depression than in the general population, which is strongly associated with poor patient-centered outcomes. Yet, depression is often not diagnosed when present, not treated when identified, and many HD patients are reluctant to accept treatment. This is likely a result of lack of high-quality evidence for the efficacy of different treatment options for comorbid depression in HD patients. OBJECTIVES Conduct an open-label, randomized controlled clinical trial among HD patients with comorbid depression to (1) compare the efficacy of an engagement interview with usual care in increasing acceptability of treatment (n=200); and (2) compare the efficacy of 12 weeks of cognitive behavioral therapy (CBT) or anti-depressant drug therapy (sertraline) for reducing the severity of depressive symptoms, and other meaningful outcomes (n=120). METHODS HD patients in up to 50 dialysis facilities in three different regions (Albuquerque, NM; Dallas, TX; Seattle, WA) will be pre-screened for the presence of clinically significant depressive symptoms. Patients with a confirmed diagnosis of major depression or dysthymia will be randomly assigned to an engagement interview or usual care to determine efficacy in increasing acceptability of treatment (n=200). Individuals who agree to treatment will be randomly assigned to individual CBT or drug therapy. CBT will be administered in a dialysis facility by a trained therapist. Sertraline will be titrated to the maximum tolerated dose using Measurement Based Care, a model of shared-decision-making. Patient-reported outcomes will be measured by a single assessor for all three sites, blinded to the treatment assignment. The primary efficacy measure will be a change in severity of depressive symptoms; secondary outcome measures will assess other important patient-reported outcomes such as somatic symptom burden, functioning, and adherence with dialysis treatment, diet, and medications. The longitudinal evolution of symptoms in patients who refuse to accept any treatment either within or outside the clinical trial will also be studied (n=40). PATIENT OUTCOMES (PROJECTED) This study will provide answers to three questions faced by HD patients with clinically significant depressive symptoms: (1) "Given my preferences, what should I expect will happen to me?"; (2) "What are my options, and what are the potential benefits and harms of these options?"; and (3) "What can I do to improve the outcomes that are most important to me?" Oversight of study will be provided by separate Patient Council and Stakeholder Council to align with PCORI's mission of generating high-integrity, evidence-based information from research guided by patients, caregivers, and broader health care community.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 21 years;
2. Undergoing thrice-weekly maintenance HD for ≥ 3 months;
3. Able to speak either English or Spanish;
4. BDI-II score ≥ 15; and
5. Meets diagnostic criteria for either current major depressive episode or dysthymia on the MINI.

Exclusion Criteria:

1. Active suicidal intent;
2. Ongoing psychotherapy or current treatment with certain anti-depressant drugs;
3. Evidence of cognitive impairment on Mini-Cog;
4. Present or past psychosis or bipolar disorder I or II on the MINI;
5. Alcohol or substance abuse diagnosed on the MINI or history of such abuse in the past three months;
6. Life expectancy < 3 months, in the judgment of the site principal investigator;
7. Anticipated to receive living related donor kidney transplantation within 3 months;
8. Pregnancy, or lactation, or women of childbearing age not willing to use adequate birth control;
9. Clinical and/or laboratory evidence of chronic liver disease;
10. History of significant active bleeding in the past three months, such as hospitalization for gastrointestinal bleeding;
11. Current use of class I anti-arrhythmic medications (e.g., propafenone, flecainide), pimozide, monoamine oxidase inhibitors, reserpine, guanethidine, cimetidine, tri-cyclic anti-depressants, triptans, tramadol, linezolid, tryptophan, and St. John's wort; and
12. Known hypersensitivity to sertraline.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2015-03-23 (Actual); Primary Completion 2017-11-15 (Actual); Study Completion 2017-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rajnish Mehrotra, MD, Principal Investigator — University of Washington
Locations (3):
- United States (3):
  - University of New Mexico, Albuquerque, New Mexico
  - University of Texas Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington

REFERENCES:
- [Background] Davison SN, Jhangri GS. The impact of chronic pain on depression, sleep, and the desire to withdraw from dialysis in hemodialysis patients. J Pain Symptom Manage. 2005 Nov;30(5):465-73. doi: 10.1016/j.jpainsymman.2005.05.013. PMID 16310620
- [Background] Weisbord SD, Fried LF, Arnold RM, Fine MJ, Levenson DJ, Peterson RA, Switzer GE. Prevalence, severity, and importance of physical and emotional symptoms in chronic hemodialysis patients. J Am Soc Nephrol. 2005 Aug;16(8):2487-94. doi: 10.1681/ASN.2005020157. Epub 2005 Jun 23. PMID 15975996
- [Background] Hedayati SS, Bosworth HB, Kuchibhatla M, Kimmel PL, Szczech LA. The predictive value of self-report scales compared with physician diagnosis of depression in hemodialysis patients. Kidney Int. 2006 May;69(9):1662-8. doi: 10.1038/sj.ki.5000308. PMID 16598203
- [Background] Kimmel PL, Peterson RA, Weihs KL, Simmens SJ, Alleyne S, Cruz I, Veis JH. Multiple measurements of depression predict mortality in a longitudinal study of chronic hemodialysis outpatients. Kidney Int. 2000 May;57(5):2093-8. doi: 10.1046/j.1523-1755.2000.00059.x. PMID 10792629
- [Background] Hedayati SS, Bosworth HB, Briley LP, Sloane RJ, Pieper CF, Kimmel PL, Szczech LA. Death or hospitalization of patients on chronic hemodialysis is associated with a physician-based diagnosis of depression. Kidney Int. 2008 Oct;74(7):930-6. doi: 10.1038/ki.2008.311. Epub 2008 Jun 25. PMID 18580856
- [Background] System, U.S.R.D., US Department of Public Health and Human Services, Public Health Service, National Institutes of Health, Bethesda, 2012.
- [Background] Glassman AH, O'Connor CM, Califf RM, Swedberg K, Schwartz P, Bigger JT Jr, Krishnan KR, van Zyl LT, Swenson JR, Finkel MS, Landau C, Shapiro PA, Pepine CJ, Mardekian J, Harrison WM, Barton D, Mclvor M; Sertraline Antidepressant Heart Attack Randomized Trial (SADHEART) Group. Sertraline treatment of major depression in patients with acute MI or unstable angina. JAMA. 2002 Aug 14;288(6):701-9. doi: 10.1001/jama.288.6.701. PMID 12169073
- [Background] Cukor D, Rosenthal DS, Jindal RM, Brown CD, Kimmel PL. Depression is an important contributor to low medication adherence in hemodialyzed patients and transplant recipients. Kidney Int. 2009 Jun;75(11):1223-1229. doi: 10.1038/ki.2009.51. Epub 2009 Feb 25. PMID 19242502
- [Background] Kutner NG, Zhang R, McClellan WM, Cole SA. Psychosocial predictors of non-compliance in haemodialysis and peritoneal dialysis patients. Nephrol Dial Transplant. 2002 Jan;17(1):93-9. doi: 10.1093/ndt/17.1.93. PMID 11773470
- [Background] Weisbord SD, Fried LF, Mor MK, Resnick AL, Unruh ML, Palevsky PM, Levenson DJ, Cooksey SH, Fine MJ, Kimmel PL, Arnold RM. Renal provider recognition of symptoms in patients on maintenance hemodialysis. Clin J Am Soc Nephrol. 2007 Sep;2(5):960-7. doi: 10.2215/CJN.00990207. Epub 2007 Aug 8. PMID 17702730
- [Background] Cukor D, Ver Halen N, Asher DR, Coplan JD, Weedon J, Wyka KE, Saggi SJ, Kimmel PL. Psychosocial intervention improves depression, quality of life, and fluid adherence in hemodialysis. J Am Soc Nephrol. 2014 Jan;25(1):196-206. doi: 10.1681/ASN.2012111134. Epub 2013 Oct 10. PMID 24115478
- [Background] Duarte PS, Miyazaki MC, Blay SL, Sesso R. Cognitive-behavioral group therapy is an effective treatment for major depression in hemodialysis patients. Kidney Int. 2009 Aug;76(4):414-21. doi: 10.1038/ki.2009.156. Epub 2009 May 20. PMID 19455196
- [Background] Atalay H, Solak Y, Biyik M, Biyik Z, Yeksan M, Uguz F, Guney I, Tonbul HZ, Turk S. Sertraline treatment is associated with an improvement in depression and health-related quality of life in chronic peritoneal dialysis patients. Int Urol Nephrol. 2010 Jun;42(2):527-36. doi: 10.1007/s11255-009-9686-y. Epub 2009 Dec 2. PMID 19953347
- [Background] Cukor D, Coplan J, Brown C, Peterson RA, Kimmel PL. Course of depression and anxiety diagnosis in patients treated with hemodialysis: a 16-month follow-up. Clin J Am Soc Nephrol. 2008 Nov;3(6):1752-8. doi: 10.2215/CJN.01120308. Epub 2008 Aug 6. PMID 18684897
- [Background] Hedayati SS, Minhajuddin AT, Toto RD, Morris DW, Rush AJ. Validation of depression screening scales in patients with CKD. Am J Kidney Dis. 2009 Sep;54(3):433-9. doi: 10.1053/j.ajkd.2009.03.016. Epub 2009 Jun 3. PMID 19493600
- [Background] Wisniewski SR, Rush AJ, Balasubramani GK, Trivedi MH, Nierenberg AA; STARD Investigators. Self-rated global measure of the frequency, intensity, and burden of side effects. J Psychiatr Pract. 2006 Mar;12(2):71-9. doi: 10.1097/00131746-200603000-00002. PMID 16728903
- [Background] Rush AJ, Trivedi MH, Ibrahim HM, Carmody TJ, Arnow B, Klein DN, Markowitz JC, Ninan PT, Kornstein S, Manber R, Thase ME, Kocsis JH, Keller MB. The 16-Item Quick Inventory of Depressive Symptomatology (QIDS), clinician rating (QIDS-C), and self-report (QIDS-SR): a psychometric evaluation in patients with chronic major depression. Biol Psychiatry. 2003 Sep 1;54(5):573-83. doi: 10.1016/s0006-3223(02)01866-8. PMID 12946886
- [Derived] Natale P, Ju A, Strippoli GF, Craig JC, Saglimbene VM, Unruh ML, Stallone G, Jaure A. Interventions for fatigue in people with kidney failure requiring dialysis. Cochrane Database Syst Rev. 2023 Aug 31;8(8):CD013074. doi: 10.1002/14651858.CD013074.pub2. PMID 37651553
- [Derived] Mehrotra R, Cukor D, Unruh M, Rue T, Heagerty P, Cohen SD, Dember LM, Diaz-Linhart Y, Dubovsky A, Greene T, Grote N, Kutner N, Trivedi MH, Quinn DK, Ver Halen N, Weisbord SD, Young BA, Kimmel PL, Hedayati SS. Comparative Efficacy of Therapies for Treatment of Depression for Patients Undergoing Maintenance Hemodialysis: A Randomized Clinical Trial. Ann Intern Med. 2019 Mar 19;170(6):369-379. doi: 10.7326/M18-2229. Epub 2019 Feb 26. PMID 30802897
- [Derived] Hedayati SS, Daniel DM, Cohen S, Comstock B, Cukor D, Diaz-Linhart Y, Dember LM, Dubovsky A, Greene T, Grote N, Heagerty P, Katon W, Kimmel PL, Kutner N, Linke L, Quinn D, Rue T, Trivedi MH, Unruh M, Weisbord S, Young BA, Mehrotra R. Rationale and design of A Trial of Sertraline vs. Cognitive Behavioral Therapy for End-stage Renal Disease Patients with Depression (ASCEND). Contemp Clin Trials. 2016 Mar;47:1-11. doi: 10.1016/j.cct.2015.11.020. Epub 2015 Nov 24. PMID 26621218
- See also: Kidney Research Institute — http://kri.washington.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants screened at 3 sites in the United States.
Groups:
- Engagement Interview: An Engagement Interview is a one-on-one session with the participant, during which a trained cognitive behavioral therapist explores barriers to treatment, including watching a 40-minute DVD together, in the dialysis facility. The DVD is given to the participant to take home.
- Control Visit: A control visit is a follow up discussion with the participant at the dialysis facility by research staff. During this visit, participants are informed of the diagnosis of major depression or dysthymia, the options for treatment available through the clinical trial, and alternatives should they decline participation in the clinical trial.
- Cognitive Behavioral Therapy: Cognitive Behavioral Therapy (CBT) consists of 10 CBT sessions of 60 minutes each, by a trained therapist in the dialysis facility (8 weekly sessions; then every other week x 2). The CBT is administered while the patient is undergoing hemodialysis unless alternative arrangements preferred by participant. During the course of intervention, study subjects undergo assessment of severity of depressive symptoms using Quick Inventory of Depressive Symptoms - Self-Report (QIDS-SR) every two weeks for the first six weeks (weeks 0, 2, 4, and 6) and every three weeks for the next six weeks (weeks 9 and 12).
- Antidepressant Drug Therapy: Anti-Depressant Drug Therapy is sertraline, a selective serotonin reuptake inhibitor, and is delivered for 12 weeks. The site investigators prescribe sertraline drug at a starting dose of 25 mg oral tablets. Dose titration is implemented using standardized assessments of depressive symptoms and drug side effects; and the research team and the patient make joint decisions to maintain, increase, or decrease the dose. This protocol establishes the highest effective but tolerable dose tailored for each patient. The QIDS-SR scale will be used to assess the clinical response for dose titration. The Frequency, Intensity, and Burden of Side Effects Ratings (FIBSER) scale will be used to assess side effects and the degree to which they interfere with day-to-day functions. The participant-specific dose at week 6, up to a maximum of 200 mg/d, will be continued for the remaining 6 weeks.
- Observational Cohort: Subjects who (1) are not willing to be randomized to study treatment and (2) do not find treatment acceptable even outside the study will be invited to participate in the prospective observational cohort for serial assessment of depressive symptoms.These subjects will only undergo assessment of severity of depressive symptoms at weeks 0, 6, and 12 using QIDS-C.
Period: Screening Intervention
Arm/Group | Engagement Interview | Control Visit | Cognitive Behavioral Therapy | Antidepressant Drug Therapy | Observational Cohort
Started | 92 (90 completed engagement interview) | 92 (89 completed control visit) | 0 | 0 | 0
Completed | 86 | 84 | 0 | 0 | 0
Not Completed | 6 | 8 | 0 | 0 | 0
Not completed — Death | 0 | 2 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0
Not completed — Determined Ineligible | 5 | 6 | 0 | 0 | 0
Period: Comparative Efficacy Trial / Observation
Arm/Group | Engagement Interview | Control Visit | Cognitive Behavioral Therapy | Antidepressant Drug Therapy | Observational Cohort
Started | 0 (Participants enrolled in screening intervention enrolled in comparative efficacy trial) | 0 (Participants enrolled in screening intervention enrolled in comparative efficacy trial) | 60 (44 completed treatment) | 60 (47 completed treatment) | 20
Completed | 0 | 0 | 55 | 58 | 18
Not Completed | 0 | 0 | 5 | 2 | 2
Not completed — Death | 0 | 0 | 2 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 2 | 2 | 2
Not completed — Administrative Withdrawal | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants in the comparitive efficacy/observation period (N=140) are a subset of participants in the screening intervention period (N=184). Total enrolled in the study is 184 (NOT 324).
Groups:
- Cognitive Behavioral Therapy: Cognitive Behavioral Therapy (CBT) consists of 10 CBT sessions of 60 minutes each, by a trained therapist in the dialysis facility (8 weekly sessions; then every other week x 2).
- Antidepressant Drug Therapy: Anti-Depressant Drug Therapy is sertraline, a selective serotonin reuptake inhibitor, and is delivered for 12 weeks. The site investigators prescribe sertraline drug at a starting dose of 25 mg oral tablets. Dose titration is implemented using standardized assessments of depressive symptoms and drug side effects.
- Obsevational Cohort: Subjects who (1) are not willing to be randomized to study treatment and (2) do not find treatment acceptable even outside the study.
- Total: Total of all reporting groups
Arm/Group | Engagement Interview | Control Visit | Cognitive Behavioral Therapy | Antidepressant Drug Therapy | Obsevational Cohort | Total
Number analyzed (Participants) | 92 | 92 | 60 | 60 | 20 | 324
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Screening Intervention Period
  years
    number analyzed (Participants) | 92 | 92 | 0 | 0 | 0 | 184
    (all) | 52 (14) | 53 (12) |  |  |  | 53 (13)
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Comparative Efficacy Trial / Observation Period
  years
    number analyzed (Participants) | 0 | 0 | 60 | 60 | 20 | 140
    (all) |  |  | 50 (13) | 53 (12) | 53 (13) | 52 (13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Screening Intervention Period
  Participants
    number analyzed (Participants) | 92 | 92 | 0 | 0 | 0 | 184
    Female | 42 | 35 |  |  |  | 77
    Male | 50 | 57 |  |  |  | 107
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Comparative Efficacy Trial / Observation Period
  Participants
    number analyzed (Participants) | 0 | 0 | 60 | 60 | 20 | 140
    Female |  |  | 27 | 25 | 7 | 59
    Male |  |  | 33 | 35 | 13 | 81
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Screening Intervention Period
  Participants
    number analyzed (Participants) | 92 | 92 | 0 | 0 | 0 | 184
    Hispanic or Latino | 27 | 22 |  |  |  | 49
    Not Hispanic or Latino | 65 | 69 |  |  |  | 134
    Unknown or Not Reported | 0 | 1 |  |  |  | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Comparative Efficacy Trial / Observation Period
  Participants
    number analyzed (Participants) | 0 | 0 | 60 | 60 | 20 | 140
    Hispanic or Latino |  |  | 14 | 20 | 5 | 39
    Not Hispanic or Latino |  |  | 46 | 39 | 15 | 100
    Unknown or Not Reported |  |  | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Screening Intervention Period
  Participants
    number analyzed (Participants) | 92 | 92 | 0 | 0 | 0 | 184
    American Indian or Alaska Native | 7 | 8 |  |  |  | 15
    Asian | 2 | 5 |  |  |  | 7
    Native Hawaiian or Other Pacific Islander | 3 | 3 |  |  |  | 6
    Black or African American | 21 | 32 |  |  |  | 53
    White | 48 | 29 |  |  |  | 77
    More than one race | 2 | 3 |  |  |  | 5
    Unknown or Not Reported | 9 | 12 |  |  |  | 21
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Comparative Efficacy Trial / Observation Period
  Participants
    number analyzed (Participants) | 0 | 0 | 60 | 60 | 20 | 140
    American Indian or Alaska Native |  |  | 3 | 6 | 1 | 10
    Asian |  |  | 1 | 2 | 3 | 6
    Native Hawaiian or Other Pacific Islander |  |  | 4 | 0 | 0 | 4
    Black or African American |  |  | 19 | 15 | 6 | 40
    White |  |  | 24 | 28 | 8 | 60
    More than one race |  |  | 2 | 0 | 2 | 4
    Unknown or Not Reported |  |  | 7 | 9 | 0 | 16
Dialysis Vintage [Median (Inter-Quartile Range); unit: months] — Months since most recent initiation of dialysis Population: Screening Intervention Period
  months
    number analyzed (Participants) | 92 | 92 | 0 | 0 | 0 | 184
    (all) | 32 [17 to 60] | 28 [15 to 78] |  |  |  | 31 [15 to 70]
Dialysis Vintage [Median (Inter-Quartile Range); unit: months] — Months since most recent initiation of dialysis Population: Comparative Efficacy Trial / Observation Period
  months
    number analyzed (Participants) | 0 | 0 | 60 | 60 | 20 | 140
    (all) |  |  | 30 [16 to 69] | 32 [18 to 61] | 21 [11 to 63] | 31 [15 to 70]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Initiated Depression Treatment
Description: The primary measure of efficacy of the Engagement Interview will be the number of patients undergoing hemodialysis with co-morbid depression who initiate treatment for the condition.
  This will be defined as one of the following:
  * Completing at least one psychotherapy session either as a part of the clinical trial or in the community within four weeks of establishing a diagnosis of major depression and/or dysthymia.
  * Receiving a supply of anti-depressant drug either as a part of the clinical trial or the treating physician within four weeks of establishing a diagnosis of major depression and/or dysthymia.
Time Frame: within four weeks of engagement interview or control visit
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement Interview | Control Visit
Number analyzed (Participants) | 86 | 84
Participants | 57 | 54
Statistical Analysis 1: Comparison: Engagement Interview vs Control Visit; Test type: Superiority; p = 0.77, Likelihood Ratio Test — a priori threshold for significance is 0.05; Likelihood ratio test obtained from logistic regression analysis adjusting for site

2. Primary Outcome: QIDS-C Score
Description: The Quick Inventory of Depressive Symptomatology Clinician-rated (QIDS-C) scale ranges from 0-27, higher scores indicate worse depression. The primary measure of efficacy of Intervention will be the mean difference in QIDS-C score at Week 12 between treatment groups.
Time Frame: Week 12 of treatment
Population: QIDS-C in Observational Cohort arm provided only for descriptive purposes, not a primary outcome.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Cognitive Behavioral Therapy: The subjects will be randomly assigned to individual CBT or sertraline drug therapy using block randomization.
  Individuals will undergo 10 CBT sessions of 60 minutes each, by a trained therapist in the dialysis facility (8 weekly sessions; then every other week x 2). The CBT will be administered while the patient is undergoing hemodialysis; however, alternative arrangements will be made upon individual patient's preferences.
  Cognitive Behavioral Therapy: Cognitive Behavioral Therapy (CBT) is a short-term psychotherapy that will focus on how the individual is thinking, behaving, and communicating today rather than on their childhood experience. The therapist will assist the patient in identifying specific distortions (cognitive assessment) and biases in thinking and will provide guidance on how to change this thinking.
- Antidepressant Drug Therapy: The subjects will be randomly assigned to individual CBT or sertraline drug therapy using block randomization. Anti-Depressant Drug Therapy will be delivered with sertraline, a selective serotonin reuptake inhibitor, and the dose will be titrated using the Measurement Based Care Protocol.
  Antidepressant Drug Therapy: The site investigators will prescribe sertraline drug at a starting dose of 25 mg oral tablets. Dose titration will be implemented using standardized assessments of depressive symptoms and drug side effects; and the research team and the patient make joint decisions to maintain, increase, or decrease the dose. This will help establish the highest effective but tolerable dose tailored for each patient. The QIDS-SR scale will be used to assess the clinical response for dose titration. The FIBSER scale will be used to assess side effects and the degree to which they interfere with day-to-day functions. The participant-specific dose at week 6, up to a maximum of 200 mg/d,
- Observational Cohort: Participants not accepting treatment but consented to be followed.
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy | Observational Cohort
Number analyzed (Participants) | 55 | 58 | 18
score on a scale | 8.1 [6.7 to 9.4] | 5.9 [4.8 to 7.1] | 7.9 [6.1 to 9.8]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; All participants randomized to treatment (N=120) were included in the pre-specified longitudinal model of QIDS-C used to estimate comparative treatment effect at 12 weeks (primary outcome). The model adjustment for clinical site and included baseline, 6 week and 12 week QIDS-C scores. Week 0 (baseline) and week 6 measurements are not pre-specified primary or secondary outcomes. The Observational Cohort arm was not included in the analysis; Test type: Superiority; p = 0.035, Wald Test — a priori threshold for significance is 0.05; The Wald test is for the week 12 comparative treatment effect from a longitudinal model of QIDS-C adjusting for clinical site; Mean Difference (Final Values) = -1.84, 95% CI 2-sided [-3.54 to -0.13] — The week 12 mean difference estimated from the longitudinal model is the difference between antidepressant drug therapy (drug) and the cognitive behavioral therapy (CBT) at 12 weeks, (drug - CBT)

3. Secondary Outcome: Number of Participants Who Accepted Depression Treatment
Description: The secondary measure of efficacy of the Engagement Interview will be the % of patients undergoing hemodialysis with co-morbid depression who are willing to accept treatment.
  This will be measured by the patient's intent and will be defined as one of the following:
  * Signing the informed consent to be randomly assigned to individual CBT or drug therapy
  * Receiving a referral by the research team and/or primary care physician and/or treating nephrologist to a therapist for psychotherapy in the community.
  * Receiving a prescription for anti-depressant drug therapy from primary care physician and/or treating nephrologist within two weeks of establishing a diagnosis of major depression/dysthymia.
Time Frame: within two weeks of engagement interview or control visit
Population: Screening Intervention Period. Two participants who died both consented to treatment within the clinical trial and therefore were counted as non-missing for accepting treatment outcome by definition even though they did not complete the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Engagement Interview | Control Visit
Number analyzed (Participants) | 86 | 86
Participants | 70 | 70
Statistical Analysis 1: Comparison: Engagement Interview vs Control Visit; Test type: Superiority; p = 0.96, Likelihood Ratio Test — a priori threshold for significance is 0.05; Likelihood Ratio Test from logistic regression analysis adjusting for clinical site

4. Secondary Outcome: BDI-II
Description: Beck Depression Inventory-II, range 0-63, higher scores indicate worse depression
Time Frame: Week 12
Population: Due to patient preference, 2 participants in the CBT arm and 5 in the Drug arm were not administered secondary outcome questionnaires at 12 weeks. In addition, due to non-response at 12 weeks, this outcome is missing for 5 participants in the CBT arm and 2 participants in the drug arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Cognitive Behavioral Therapy: The subjects will be randomly assigned to individual CBT or sertraline drug therapy using block randomization.
  Individuals will undergo 10 CBT sessions of 60 minutes each, by a trained therapist in the dialysis facility (8 weekly sessions; then every other week x 2).
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 48 | 51
score on a scale | 18.7 [15.2 to 22.2] | 14.1 [11.2 to 17.0]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Mean Difference (Final Values) = -3.7, 95% CI 2-sided [-7.4 to -0.02] — The mean difference estimate is from longitudinal model adjusted for clinical site. It is the difference in scores between treatment groups (Drug - CBT) at 12 weeks. All participants are included in the longitudinal model (N=120)

5. Secondary Outcome: GAD-7
Description: Generalized Anxiety Disorder 7-item Scale, range 0-21, higher scores indicate worse anxiety
Time Frame: Week 12
Population: Due to patient preference, 2 participants in the CBT arm and 5 in the Drug arm were not administered secondary outcome questionnaires at 12 weeks. In addition, due to non-response at 12 weeks, this outcome is missing for 3 participants in the CBT arm and 4 participants in the drug arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 50 | 49
score on a scale | 7.5 [5.9 to 9.2] | 6.5 [4.9 to 8.1]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-3.1 to 0.8] — [estimate comment as in outcome 4, analysis 1]

6. Secondary Outcome: Sheehan Disability Scale
Description: range 0-30, higher scores indicate worse disability
Time Frame: Week 12
Population: Due to patient preference, 2 participants in the CBT arm and 5 in the Drug arm were not administered secondary outcome questionnaires at 12 weeks. In addition, due to non-response at 12 weeks, this outcome is missing for 3 participants in the CBT arm and 1 participant in the drug arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 50 | 52
score on a scale | 15.2 [12.8 to 17.6] | 11.0 [8.7 to 13.3]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Mean Difference (Final Values) = -3.1, 95% CI 2-sided [-6.2 to -0.1] — [estimate comment as in outcome 4, analysis 1]

7. Secondary Outcome: SF-36 Energy/Vitality
Description: Energy/vitality subscale of the 36-Item Short Form Health Survey, range 0-100, higher scores indicate better energy/vitality
Time Frame: Week 12
Population: Due to patient preference, 2 participants in the CBT arm and 5 in the Drug arm were not administered secondary outcome questionnaires at 12 weeks. In addition, due to non-response at 12 weeks, this outcome is missing for 2 participants in the CBT arm and 4 participants in the drug arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 51 | 49
score on a scale | 39.2 [33.4 to 44.9] | 53 [45.7 to 60.3]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Mean Difference (Final Values) = 10.2, 95% CI 2-sided [1.3 to 19.0] — [estimate comment as in outcome 4, analysis 1]

8. Secondary Outcome: Global Quality of Life Scale
Description: range 0-10, higher scores indicate better quality of life
Time Frame: Week 12
Population: Due to patient preference, 2 participants in the CBT arm and 5 in the Drug arm were not administered secondary outcome questionnaires at 12 weeks.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 53 | 53
score on a scale | 5.6 [5.0 to 6.2] | 6.4 [5.8 to 7.0]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-0.2 to 1.4] — [estimate comment as in outcome 4, analysis 1]

9. Secondary Outcome: Satisfaction With Life Scale
Description: range 1-35, higher scores indicate better satisfaction
Time Frame: Week 12
Population: Due to patient preference, 2 participants in the CBT arm and 5 in the Drug arm were not administered secondary outcome questionnaires at 12 weeks. In addition, due to non-response at 12 weeks, this outcome is missing for 1 participant in the drug arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 53 | 52
score on a scale | 16.8 [14.9 to 18.6] | 20.1 [17.9 to 22.3]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Mean Difference (Final Values) = 2.6, 95% CI 2-sided [0.1 to 5.1] — [estimate comment as in outcome 4, analysis 1]

10. Secondary Outcome: Perceived Social Support
Description: Multi-Dimensional Scale of Perceived Social Support, range 1-7, higher scores indicate better social support
Time Frame: Week 12
Population: Due to patient preference, 2 participants in the CBT arm and 5 in the Drug arm were not administered secondary outcome questionnaires at 12 weeks. In addition, due to non-response at 12 weeks, this outcome is missing for 2 participants in the drug arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 53 | 51
score on a scale | 4.7 [4.3 to 5.1] | 4.6 [4.2 to 5.1]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Mean Difference (Final Values) = -0.01, 95% CI 2-sided [-0.5 to 0.5] — [estimate comment as in outcome 4, analysis 1]

11. Secondary Outcome: PSQI
Description: Pittsburgh Sleep Quality Index, range 0-21, higher scores indicate worse sleep quality
Time Frame: Week 12
Population: Due to patient preference, 2 participants in the CBT arm and 5 in the Drug arm were not administered secondary outcome questionnaires at 12 weeks. In addition, due to non-response at 12 weeks, this outcome is missing for 11 participants in the CBT arm and 13 participants in the drug arm.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 42 | 40
score on a scale | 9.5 [8.1 to 10.8] | 6.8 [5.5 to 8.1]

12. Secondary Outcome: Exercise
Description: Single item activity measure, range 1-6, higher indicates less activity
Time Frame: Week 12
Population: as for outcome 9
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 53 | 52
score on a scale | 3.5 [3.1 to 4.0] | 3.2 [2.8 to 3.7]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Mean Difference (Final Values) = 0.1, 95% CI 2-sided [-0.5 to 0.7] — [estimate comment as in outcome 4, analysis 1]

13. Secondary Outcome: Percentage of Dialysis Treatment Sessions Skipped and/or Shortened
Description: Treatment Adherence with Dialysis as defined by the percentage of all dialysis sessions skipped and/or requested by the patient to be shortened by ≥ 10 minutes over the 12-week intervention period. Dialysis sessions missed due to hospitalization will not be included as a skipped treatment.
Time Frame: Over 12 Weeks
Measure: Mean (95% Confidence Interval); unit: percentage of sessions skipped/shortened
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 55 | 58
percentage of sessions skipped/shortened | 22.2 [16.4 to 28.0] | 17.3 [13.0 to 21.6]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Risk Ratio (RR) = 0.78, 95% CI 2-sided [0.55 to 1.10] — The mean difference estimate is from a negative binomial model adjusted for clinical site. It is the rate of sessions skipped/shortened in the Drug group (numerator) compared to CBT (denominator)

14. Secondary Outcome: Percent Inter-dialytic Weight Gain
Description: Treatment Adherence with Fluid Intake as defined by inter-dialytic weight gain (as % of post-dialysis weight) during Week 12 of the study
Time Frame: Week 12
Population: In addition to participants withdrawn / died, 11 participants were missing average weight gain at week 12: 3 in CBT arm and 8 in Drug arm.
Measure: Mean (95% Confidence Interval); unit: percentage of body weight
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 52 | 50
percentage of body weight | 2.6 [2.3 to 3.0] | 2.9 [2.5 to 3.4]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.54 to 0.34] — [estimate comment as in outcome 4, analysis 1]

15. Secondary Outcome: Serum Phosphorus Level
Description: Treatment Adherence with Diet and/or Medications as defined by Serum phosphorus level measured as a part of routine clinical care during the third month of participation in the study.
Time Frame: Week 12
Population: In addition to participants withdrawn / died, 8 participants were missing serum phosphorus level at week 12: 3 in CBT arm and 5 in Drug arm.
Measure: Mean (95% Confidence Interval); unit: mg/dl
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
Number analyzed (Participants) | 52 | 53
mg/dl | 6.1 [5.6 to 6.6] | 6.3 [5.9 to 6.8]
Statistical Analysis 1: Comparison: Cognitive Behavioral Therapy vs Antidepressant Drug Therapy; Test type: Superiority; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.25 to 0.75] — [estimate comment as in outcome 4, analysis 1]

ADVERSE EVENTS:
Time Frame: Participants followed from randomization to treatment to 30 days after end of treatment period (4 months).
Description: Participants in the comparative efficacy trial (CBT-I or drug arms) were asked at each study visit if they had experienced any adverse events. Adverse events were not captured for participants in the observation arm or participants only randomized to engagement or control visit.
Arm/Group | Cognitive Behavioral Therapy | Antidepressant Drug Therapy
All-Cause Mortality (participants affected / at risk) | 2/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 11/60 | 14/60
Other Adverse Events (participants affected / at risk) | 4/60 | 12/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (N=60) | Antidepressant Drug Therapy (N=60)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0)
Afib (Cardiac disorders) | 1 (1) | 0 (0)
Syncope (Cardiac disorders) | 0 (0) | 1 (1)
Volume overload (Cardiac disorders) | 2 (2) | 2 (2)
Cardiovascular event (Cardiac disorders) | 1 (1) | 0 (0) — Fatal
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Rectal bleeding (Gastrointestinal disorders) | 0 (0) | 1 (1)
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Catheter infection (Infections and infestations) | 0 (0) | 1 (1)
Healthcare-associated pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 1 (2) | 0 (0)
Leg fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Leg amputation (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Vertigo, facial palsy (shingles) (Nervous system disorders) | 0 (0) | 1 (1)
Convulsions (Nervous system disorders) | 0 (0) | 1 (1)
Vaginal bleeding (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Kidney transplant (Surgical and medical procedures) | 0 (0) | 1 (1)
Arteriovenous grafts vascular access surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Leg ischemia (Vascular disorders) | 1 (1) | 0 (0)
Arteriovenous graft malfunction (Vascular disorders) | 0 (0) | 1 (1)
Renal artery aneurysm (Vascular disorders) | 0 (0) | 1 (1)
Unknown System Organ Class (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Participant died at home
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitive Behavioral Therapy (N=60) | Antidepressant Drug Therapy (N=60)
Dizziness (Cardiac disorders) | 0 (0) | 5 (5)
Vomiting (Gastrointestinal disorders) | 4 (4) | 6 (7)
Fatigue (General disorders) | 0 (0) | 5 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT02358343/Prot_SAP_000.pdf